CLINICAL TRIAL: NCT06621225
Title: A Randomized Trial on the Utilization of Endocuff-assisted Colonoscopy and Computer-aided Detection in Optimizing Colonoscopies in the Elderly
Brief Title: Artificial Intelligence in Colonoscopy
Acronym: AIColonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pankaj Patel (Other)
Responsible Party: Sponsor-Investigator, Pankaj Patel, Gastroenterologist and Medical Director of The Surgery and Endoscopy Center, The Surgery and Endoscopy Center of Sebring
Organization: The Surgery and Endoscopy Center of Sebring (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: Pro00069956
Record Dates: First submitted 2024-09-07; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Carcinoma
Keywords: Colonoscopy; Mucosal Exposure Device; Artificial Intelligence
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into one of three study groups: the primary intervention arm, where colonoscopy was performed using the CADe in combination with the MED; the second group underwent colonoscopy solely with the MED, while the control group underwent colonoscopy solely with the WLE. Randomization was executed by a scheduler responsible for patient appointments at the practice, ensuring impartial allocation, with the investigators maintaining no involvement in subject assignment to study arms. We used a Convolutional Neural Network-based CADe system, GI Genius, acquired for licensed use from Medtronic Inc., Minneapolis, MN. The MED employed was the EndoCuff Vision (ECV) developed by Olympus America, Center Valley, PA, which constitutes part of the standard equipment available. All detected lesions were identified and excised throughout the colonoscopy procedures, and specimens were promptly sent for histopathological analysis.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Primary Intervention Arm (Experimental): In this arm, colonoscopy was performed using Computer Aided detection in combination with a Mucosal Exposure Device, which is FDA approved.
  Interventions: Device: Artificial Intelligence; Device: Mucosal Exposure Device
- Secondary Intervention Arm (Experimental): In this arm, participants underwent colonoscopy solely with an FDA approved Mucosal Exposure Device
  Interventions: Device: Mucosal Exposure Device
- Control group (No Intervention): In this arm, the participants underwent standard white light endoscopy without any intervention.

INTERVENTIONS:
Device: Artificial Intelligence — Medtronic GI Genius is an advanced AI-powered platform designed to assist gastroenterologists during colonoscopies. Utilizing deep learning algorithms, it analyzes real-time endoscopic images to detect and highlight polyps and other abnormalities, enhancing the detection rate and accuracy. The system provides visual cues to guide physicians in identifying potentially problematic areas that might be missed by the human eye alone. This technology aims to improve diagnostic precision, reduce missed detections, and ultimately enhance patient outcomes by facilitating earlier and more accurate interventions. GI Genius integrates seamlessly with existing endoscopy equipment, offering a valuable tool in the fight against colorectal cancer.
  Arms: Primary Intervention Arm
Device: Mucosal Exposure Device — The Olympus Endocuff is an innovative device designed to enhance the effectiveness of colonoscopy procedures. It is a soft, flexible cuff that attaches to the end of the colonoscope and features multiple protruding "fingers" that help to improve mucosal exposure. By providing better visibility and maneuverability, the Endocuff helps gastroenterologists navigate and inspect the colon more thoroughly. It aids in the detection of polyps and other abnormalities by flattening folds and improving the overall view of the colon lining. This enhanced visualization contributes to more accurate diagnoses and can potentially reduce the miss rate of significant lesions, ultimately leading to better patient outcomes.
  Arms: Primary Intervention Arm; Secondary Intervention Arm

SUMMARY:
N = 264 patients (50% female) aged 75 years and above undergoing colonoscopy were enrolled. Patients were randomly assigned into one of the three intervention groups: the primary intervention arm (CADe in combination with the MED), the second group with MED alone, and the control group with WLE. All detected lesions were removed and sent to histopathology for diagnosis. The primary outcome was the adenoma detection rate. Secondary outcomes were adenoma detection in the left colon in our cohort of patients.

DETAILED DESCRIPTION:
264 patients, with an equal gender distribution (50% female), aged 75 years and above, undergoing screening and diagnostic colonoscopy at The Surgery and Endoscopy Center of Sebring, Sebring, Florida, were enrolled in this study. The eligibility criteria for a randomized controlled trial (RCT) comparing AI and mucosal exposure devices together, mucosal exposure devices alone, and white light endoscopy in patients 75 years and older could be structured as follows.

Patients were randomly allocated into one of three study groups: the primary intervention arm, where colonoscopy was performed using the CADe in combination with the MED; the second group underwent colonoscopy solely with the MED, while the control group underwent colonoscopy solely with the WLE. We used a Convolutional Neural Network-based CADe system, GI Genius, acquired for licensed use from Medtronic Inc., Minneapolis, MN. The MED employed was the EndoCuff Vision (ECV) developed by Olympus America, Center Valley, PA, which constitutes part of the standard equipment available. All detected lesions were identified and excised throughout the colonoscopy procedures, and specimens were promptly sent for histopathological analysis.

The primary outcome of interest was adenoma detection rate (ADR), defined as the percentage of patients in whom at least one histologically proven adenoma or carcinoma was identified during colonoscopy. Secondary outcomes included ADR in the left colon in our cohort of patients.

This study was conducted according to accepted ethical principles and approved by the institutional review board (IRB) of "The Surgery and Endoscopy Center of Sebring." Informed consent was obtained from all participants before enrollment, and measures were taken to ensure patient confidentiality and data protection throughout the study period.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 75 years and older.
2. Patients who were able to provide informed consent or had a legally authorized representative who can consent on their behalf.
3. Patients who were deemed fit for colonoscopy based on a pre-procedure evaluation.

Exclusion criteria

1. Patients with acute gastrointestinal conditions such as active colitis, acute diverticulitis, or bowel obstruction.
2. Patients with a history of major colorectal surgery that might alter normal colon anatomy (e.g., colectomy).
3. Patients with severe comorbid conditions that would contraindicate colonoscopy, such as severe cardiopulmonary disease or advanced liver disease.
4. Patients with uncorrected coagulopathies or those on anticoagulation therapy that cannot be safely managed around the time of the procedure.
5. Patients who are unable to adequately prepare the bowel for colonoscopy.
6. Patients who refuse to participate in the study or have a legally authorized representative who refuses consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 264 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 181 days
  The primary outcome of interest was adenoma detection rate (ADR), defined as the percentage of patients in whom at least one histologically proven adenoma or carcinoma was identified during colonoscopy.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 181 days
  Secondary outcomes included Adenoam Detection Rate in the left colon in our cohort of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj J Patel, MD, Principal Investigator — The Surgery and Endoscopy Center of Sebring
Locations (1):
- The Surgery and Endoscopy Center of Sebring, Sebring, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) might not be shared in clinical trial registration for several reasons. Firstly, sharing IPD raises privacy concerns, as de-identification processes may not fully protect participants' confidentiality. Ethical obligations to safeguard participants' sensitive health information must be upheld. Secondly, consent limitations could prevent sharing, especially if participants were not explicitly informed that their data might be shared with external parties. Additionally, proprietary concerns could restrict data sharing if the data are tied to intellectual property or are part of ongoing research. Lastly, regulatory or legal restrictions in specific regions or institutions may limit the ability to share IPD.

REFERENCES:
- [Background] Pohl H, Robertson DJ. Colorectal cancers detected after colonoscopy frequently result from missed lesions. Clin Gastroenterol Hepatol. 2010 Oct;8(10):858-64. doi: 10.1016/j.cgh.2010.06.028. Epub 2010 Jul 22. PMID 20655393
- [Background] Dekker E, Tanis PJ, Vleugels JLA, Kasi PM, Wallace MB. Colorectal cancer. Lancet. 2019 Oct 19;394(10207):1467-1480. doi: 10.1016/S0140-6736(19)32319-0. PMID 31631858